CLINICAL TRIAL: NCT04990934
Title: Transitioning Care: Perspectives of Older Women With Early Breast Cancer on Current Telemedicine Modalities
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2105
Record Dates: First submitted 2021-06-25; First posted 2021-08-05 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer Female; Breast Cancer
Keywords: Telemedicine
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Video Telemedicine: 20 participants will have used video telemedicine for appointments with their treating oncologist.
  Interventions: Behavioral: Semistructured Interview
- Telephone Telemedicine: 10 participants will have used telephone telemedicine for appointments with their treating oncologist.
  Interventions: Behavioral: Semistructured Interview

INTERVENTIONS:
Behavioral: Semistructured Interview — Patients with breast cancer (Stage I-III) will be interviewed about their experiences of telemedicine.

SUMMARY:
Explosive growth in the use of telemedicine (video or telephone visits) has followed the onset of the coronavirus disease 2019 (COVID-19) pandemic in order to meet healthcare needs while avoiding unnecessary exposure risks in ambulatory care spaces. Accordingly, in March 2020, the Centers for Medicare & Medicaid Services expanded reimbursement for telemedicine visits to equal that of in-person services. The policy and infrastructure that enabled this emergency transition is laying the groundwork for enduring expansion of elective telemedicine, a technology that could significantly decrease the burden of medical care in older patients with cancer. To benefit from telehealth, patients must have a certain level of knowledge and capacity to engage with technology, which can be a challenge for some older adults because of inexperience, access, and disability. As cancer is mainly a disease of older adults, with a median age of 65 at diagnosis for most cancer types, this is a significant limitation on the utility of telemedicine in oncology.

The goal of our study is to better understand older breast cancer patients' experiences with telephone and video telemedicine with regard to visit convenience, completeness, and interpersonal satisfaction through semi-structured interviews with patients.

DETAILED DESCRIPTION:
Methods:

30 participants will be consented in this study. 20 will have participated in video telemedicine appointments with their treating breast cancer oncologists, and 10 will have used telephone. Semi-structured interviews lasting no more than 30 minutes will be conducted to ascertain the participant's (1) reason for choosing a certain telemedicine modality, (2) perception of telemedicine visit convenience, completeness, and interpersonal satisfaction compared to in-person visits, and (3) use of peripheral virtual support from healthcare team, such as messaging in MyChart. After the interview has been conducted, the patient will be asked complete the patient-reported portion of the Geriatric Assessment (GA) either through an internet link, or verbally with the research staff reading the questions and recording the answers. Data pertaining to the participant's breast cancer diagnosis and treatment will be extracted from Epic@UNC.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 65 or older
* diagnosed with early breast cancer (Stage I-III)
* completed primary treatment (surgery, chemotherapy, radiation treatment)
* received in-person outpatient care at North Caroline Cancer Hospital before transitioning to telemedicine after March 2020
* providing written informed consent
* able to understand and speak English.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria stated above will be excluded. There will be no further exclusion criteria.

Ages: 65 Years to 110 Years | Sex: Female
Age Groups: Older Adult
Gender Based: Yes — Self-identifying women will be eligible
Study Population: Patients diagnosed with early BC (Stage I-III) who have completed primary treatment and received in-person outpatient care at North Carolina Cancer Hospital before transitioning to telemedicine after March 2020.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Qualitative Summaries of Interviews about Participant Experience with Telemedicine | 3 months post study start
  Qualitative Summaries derived from content analysis of semi-structured interview transcripts around themes and sub themes of convenience, psychosocial experience, baseline comfort with technology, preference for telephone vs. video visits, and desire to continue using telemedicine in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Buse, MM, BA, BM, Principal Investigator — UNC School of Medicine Student
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: 9 to 24 months following publication
Access Criteria: When data sharing is permitted, a Data Use Agreement (DUA) specifying the uses of such data to be shared must be in place before any data is shared. Requests can be submitted to the UNC Office of Industry Contracting for processing. The Principal Investigator must confirm that the DUA has been fully executed and IRB, IEC, or REB approval has been granted before sharing data.
URL: https://research.unc.edu/sponsored-research/resources/industry-contracting/

REFERENCES:
- [Background] Sirintrapun SJ, Lopez AM. Telemedicine in Cancer Care. Am Soc Clin Oncol Educ Book. 2018 May 23;38:540-545. doi: 10.1200/EDBK_200141. PMID 30231354
- [Background] Eberly LA, Kallan MJ, Julien HM, Haynes N, Khatana SAM, Nathan AS, Snider C, Chokshi NP, Eneanya ND, Takvorian SU, Anastos-Wallen R, Chaiyachati K, Ambrose M, O'Quinn R, Seigerman M, Goldberg LR, Leri D, Choi K, Gitelman Y, Kolansky DM, Cappola TP, Ferrari VA, Hanson CW, Deleener ME, Adusumalli S. Patient Characteristics Associated With Telemedicine Access for Primary and Specialty Ambulatory Care During the COVID-19 Pandemic. JAMA Netw Open. 2020 Dec 1;3(12):e2031640. doi: 10.1001/jamanetworkopen.2020.31640. PMID 33372974
- [Background] Narasimha S, Madathil KC, Agnisarman S, Rogers H, Welch B, Ashok A, Nair A, McElligott J. Designing Telemedicine Systems for Geriatric Patients: A Review of the Usability Studies. Telemed J E Health. 2017 Jun;23(6):459-472. doi: 10.1089/tmj.2016.0178. Epub 2016 Nov 22. PMID 27875667
- [Background] Rowland JH, Bellizzi KM. Cancer survivorship issues: life after treatment and implications for an aging population. J Clin Oncol. 2014 Aug 20;32(24):2662-8. doi: 10.1200/JCO.2014.55.8361. Epub 2014 Jul 28. PMID 25071099
- See also: Coronavirus Preparedness and Response Supplemental Appropriations Act, 2020, HR 6074, 116th Cong (2020) — https://www.govtrack.us/congress/bills/116/hr6074
- See also: Medicare and Medicaid Programs, Basic Health Program, and Exchanges; Additional Policy and Regulatory Revisions in Response to the COVID-19 Public Health Emergency — https://www.federalregister.gov/documents/2020/05/08/2020-09608/medicare-and-medicaid-programs-basic-health-program-and-exchanges-additional-policy-and-regulatory
- See also: Final Policy, Payment, and Quality Provisions Changes to the Medicare Physician Fee Schedule for Calendar Year 2021 (December 1, 2020). — https://www.cms.gov/newsroom/fact-sheets/final-policy-payment-and-quality-provisions-changes-medicare-physician-fee-schedule-calendar-year-1
- See also: Pew Research Center: Tech Adoption Climbs Among Older Adults — https://www.pewresearch.org/internet/2017/05/17/technology-use-among-seniors/